CLINICAL TRIAL: NCT07002242
Title: A Clinical Study of the Interactions Between Azvudine Tablets (FNC) and Aluvia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GQ-FNC-108
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Azvudine
MeSH Terms: interventions — lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : FNC+ Aluvia;Aluvia;FNC (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Aluvia; Drug: Azvudine tablets(FNC); Drug: Aluvia
- Group 2 : FNC;FNC+Aluvia;Aluvia (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Aluvia; Drug: Azvudine tablets(FNC); Drug: Aluvia
- Group 3 : Aluvia;FNC;FNC+Aluvia (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Aluvia; Drug: Azvudine tablets(FNC); Drug: Aluvia

INTERVENTIONS:
Drug: Azvudine tablets(FNC) and Aluvia — FNC 3 mg each time, 1 time a day, orally, for 5 consecutive days. Aluvia(Lopinavir / Ritonavir tablets): 400 mg/100 mg (2 tablets) each time, 2 time a day, orally, for 5 consecutive days.
Drug: Azvudine tablets(FNC) — FNC: 3 mg each time, 1 time a day, orally, for 5 consecutive days
Drug: Aluvia — Aluvia(Lopinavir / Ritonavir tablets): 400 mg/100 mg (2 tablets) each time, 2 time a day, orally, for 5 consecutive days.

SUMMARY:
Azvudine(FNC)，a nucleoside reverse transcriptase inhibitor, make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance. FNC is a broad-spectrum RNA virus inhibitor that inhibits the novel coronavirus RNA-dependent RNA polymerase (RdRp).

This is a clinical study to evaluate the Interactions between Azvudine Tablets (FNC) and Aluvia in healthy subjects. This is a single-center, randomized, open-label, three-cycles, three-treatment crossover clinical trial. Subjects was administered orally for 5 consecutive days each cycle, and the washout period between each cycle was 7 days. Biological sample collection and safety examination were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged ≥ 18 years old and ≤ 45 years old, regardless of gender;
2. Body mass index (BMI) within the range of 19.0-26.0 (including the critical value) (BMI = weight (kg) / height 2 (m2)), the weight of men should be ≥ 50.0kg, and the weight of women should be ≥ 45.0kg;
3. Those who had no birth plan within 2 weeks before screening and within 6 months after the end of the trial and agree to take effective non-drug contraceptive measures during the trial;
4. Understand and sign the informed consent form.

Exclusion Criteria:

1. Persons with allergic constitutions, history of drug or food allergies, especially those who were allergic to any ingredient in this product and its excipients;
2. Individuals with a history of hypoglycemia;
3. Individuals deemed ineligible by the clinical research physician due to significant clinical abnormalities in medical history, physical examination, laboratory tests, and other related examinations;
4. Individuals with a history of smoking addiction within 12 months prior to screening (the number of cigarettes smoked ≥5 per day);
5. Individuals with a history of alcohol abuse within the past 12 months (consuming ≥14 units of alcohol weekly: 1 unit = 285 mL of beer, or 25 mL of spirits, or 150 mL of wine), or who tested positive for alcohol on breath tests prior to study enrollment (testing value >0mg/100mL);
6. Individuals with a history of substance abuse within the past 12 months or who tested positive for addictive substances prior to enrollment;
7. Individuals who underwent surgery within the past 3 months, especially those who had had surgeries that would affect drug absorption, distribution, metabolism, or excretion, or those planning to undergo surgery during the study;
8. Individuals who had taken any medication that interacts with the trial drug in the 30 days prior to screening, such as strong CYP3A inhibitors (e.g., clarithromycin, indinavir, itraconazole, etc.);
9. Individuals with a history of cardiovascular, liver, kidney, pulmonary, gastrointestinal, neurological diseases, especially any surgical conditions or disorders that might affect drug absorption, distribution, metabolism, and excretion, or any surgical conditions or disorders that might pose hazards to participants;
10. Individuals with febrile illness within the 3 days prior to screening;
11. Individuals who had participated in any other clinical trials within the past 3 months;
12. Individuals with any history of prescription drugs, over-the-counter drugs, herbal medicine, or dietary supplements within 14 days prior to screening;
13. Individuals who had been vaccinated against the novel coronavirus within 14 days before screening or other vaccines within 3 months before screening or planed to be vaccinated during the trial;
14. Individuals who had consumed excessive tea, coffee, and/or caffeinated, xanthine, or alcoholic beverages (more than 8 cups, 1 cup = 250 mL) daily within the 3 months prior to screening;
15. Individuals who had lost blood or donated ≥200 mL within the past 8 weeks;
16. Pregnant or breastfeeding women;
17. Individuals who could not tolerate venipuncture or had a history of vasovagal syncope;
18. Individuals deemed unsuitable for this study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration at Steady State (Cmax, ss) of Azvudine, Lopinavir and Ritonavir | Blood samples were collected on Day 3, 4, 5, 14, 15, 16, 25, 26 and 27 of the study.
Pharmacokinetics (PK): Time to Maximum Plasma Concentration at Steady State (Tmax, ss) of Azvudine, Lopinavir and Ritonavir | Blood samples were collected on Day 3, 4, 5, 14, 15, 16, 25, 26 and 27 of the study.
Pharmacokinetics (PK): Elimination of Terminal Half-Life (t1/2) of Azvudine, Lopinavir and Ritonavir | Blood samples were collected on Day 3, 4, 5, 14, 15, 16, 25, 26 and 27 of the study.

SECONDARY OUTCOMES:
Occurrence of Adverse Events | From enrollment to the end of the study on Day 28.
  Clinical presentation characteristics, severity, onset time, duration of adverse events, management measures, outcomes, and the correlation with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin People's Hospital, Tianjin, China